CLINICAL TRIAL: NCT06678620
Title: A Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of a 24-valent Pneumococcal Polysaccharide Conjugate Vaccine in People Aged 18 Years and Older
Brief Title: Phase II Clinical Trial of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Reinovax Biologics Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT183
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): 248 participants will be randomized to receive Reinovax PCV24 formulation 1. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: Reinovax PCV24 formulation 1
- Experimental group 2 (Experimental): 248 participants will be randomized to receive Reinovax PCV24 formulation 2. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: Reinovax PCV24 formulation 2
- Experimental group 3 (Experimental): 248 participants will be randomized to receive Reinovax PCV24 formulation 3. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: Reinovax PCV24 formulation 3
- Active control group (Active Comparator): 248 participants will be randomized to receive PPSV23. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: Reinovax PCV24 formulation 1 — One dose of Reinovax PCV24 formulation 1（0.5mL）
  Arms: Experimental group 1
Biological: Reinovax PCV24 formulation 2 — One dose of Reinovax PCV24 formulation 1（0.5mL）
  Arms: Experimental group 2
Biological: Reinovax PCV24 formulation 3 — One dose of Reinovax PCV24 formulation 1（0.5mL）
  Arms: Experimental group 3
Biological: PPSV23 — One dose of PPSV23 (0.5 mL) contains 1、2、3、4、5、6B、7F、8、9N、9V、10A、11A、12F、14、15B、17F、18C、19A、19F、20、22F、23F and33F saccharides.
  Arms: Active control group

SUMMARY:
A phase II clinical trial of a 24-valent pneumococcal conjugate vaccine (PCV24) developed by Shanghai Reinovax Biologics Co., LTD will be conducted in Chinese adults aged 18 years and older. The study's objective is to evaluate the safety and immunogenicity of PCV24. The trial is a single-center, randomized, blinded, parallel-controlled, non-inferiority design II clinical trial.

DETAILED DESCRIPTION:
Phase II clinical trial of the 24-valent pneumococcal conjugate vaccine (PCV24) developed by Shanghai Reinovax Biologics Co., LTD will be conducted in Chinese adults aged 18 years and older. The study's objective is to evaluate the safety and immunogenicity of PCV24. The active control vaccine is a 23-valent pneumococcal polysaccharide vaccine (23-valent pneumococcal polysaccharide vaccine, PPSV23) produced by the Chengdu Institute of Biological Products.

At least 992 participants will be enrolled, including 496 adults aged 18-60 and 496 elderly people aged ≥61. Participants will be randomized 1:1:1:1 to receive one dose of PCV24 formulation 1, PCV24 formulation 2, PCV24 formulation 3,or PPSV23.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers aged 18 and above on the day of screening, and can provide legal identification;
2. Informed consent must be obtained from the volunteer and signed informed consent form;
3. Volunteers are able and willing to comply with the requirements of the clinical trial protocol and can attend all visits;
4. Armpit body temperature ≤ 37.0 °C on the day of enrollment.

   Exclusion Criteria:
5. Previous vaccination with pneumococcal conjugate vaccine, prior vaccination with pneumococcal polysaccharide vaccine for less than 3 years, or previous history of invasive disease caused by Streptococcus pneumoniae;
6. Have any history of severe allergies in the past, such as anaphylactic shock, allergic laryngeal edema, Henoch-Schonlein purpura, thrombocytopenic purpura, local allergic necrosis reaction (Athus reaction), etc.;
7. Have been diagnosed with congenital or acquired immunodeficiency, or have recently received immunosuppressant therapy, such as systemic glucocorticoid therapy such as prednisone or similar drugs >5 mg/day for more than 2 consecutive weeks in 1 month prior to vaccination);
8. Suffering from more serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension that cannot be controlled by medication (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg when measured on site);
9. Those who have acute febrile illness or acute infectious disease or have cold symptoms, advanced influenza and take medication;
10. History of nervous system damage, severe congenital malformations, severe developmental disorders, severe genetic defects, severe malnutrition, etc.;
11. Have a history or family history of epilepsy, encephalopathy, or psychiatric disorders;
12. Those who have been diagnosed with thrombocytopenia, any abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities, etc.) or contraindications to intramuscular injection such as anticoagulant therapy;
13. asplenia, functional asplenia, and asplenia or splenectomy due to any cause;
14. Suffering from severe chronic diseases or the disease is in the advanced stage and cannot be controlled smoothly;
15. Have received blood or blood-related products or immunoglobulins within 3 months;
16. Received live attenuated vaccine within 14 days;
17. Other vaccinations within 7 days;
18. Received other investigational drugs or vaccines within 1 month;
19. Is participating in or plans to participate in clinical studies of other drugs or vaccines during the study period;
20. Any other condition that, in the opinion of the investigator, may interfere with the study evaluation;
21. Exclusion Criteria for Partial Populations:

Females of childbearing potential (18~49 years old): positive urine pregnancy test on the day of enrollment, lactation, or pregnancy plans within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 992 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | 0~30 days after vaccination
  The incidence of adverse events within 30 days after vaccination.
Incidence of serious adverse events (SAE) | 0-6 months after vaccination
  Incidence of SAE during the period of safety monitoring
Positive conversion rate of specific IgG antibodies by serotype | 0~30 days after vaccination
  The positive conversion rate of IgG antibody of each serotype covered by pneumococcal vaccine detected by Enzyme linked immunosorbent assay (ELISA) 30 days after immunization in each group.

SECONDARY OUTCOMES:
The geometric mean concentration (GMC) of specific IgG antibodies detected by ELISA of each serotype of pneumococcus | 0~30 days after vaccination
  The geometric mean concentration (GMC) of specific IgG antibodies detected by ELISA of each serotype of pneumococcus in subjects 30 days after immunization in each group

OTHER OUTCOMES:
the exploratory subgroup, the geometric mean concentration (GMT) of the pneumococcal vaccine was covered by multiplexed opsonophagocytic assay (MOPA) | 0~30 days after vaccination
  In the exploratory subgroup, the geometric mean concentration (GMT) of the pneumococcal vaccine was covered by multiplexed opsonophagocytic assay (MOPA) 30 days before and 30 days after immunization.
Exploratory subgroup, pneumococcal vaccine coverage of all serotypes/partial serotypes IgG and/or sIgA antibody levels in saliva | before vaccination, 30 days, and 6 months after vaccination
  Exploratory subgroup, pneumococcal vaccine coverage of all serotypes/partial serotypes IgG and/or sIgA antibody levels in saliva before vaccination, 30 days, and 6 months after vaccination
Exploratory subgroup, pneumococcal colonization in the nasopharynx of subjects | before vaccination, 30 days, and 6 months after vaccination.
  Exploratory subgroup, pneumococcal colonization in the nasopharynx of subjects before vaccination, 30 days, and 6 months after vaccination.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Pizhou Center for Disease Control and Prevention, Pizhou, Jiangsu
  - Xuzhou Center for Disease Control and Prevention, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No